CLINICAL TRIAL: NCT05117073
Title: Risk Factors of Spontaneous Fungal Peritonitis in Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdelrhman, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-10-53
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Spontanous Fungal Peritonitis
Keywords: spontanous fungal peritonitis, liver cirrhosis, risk factors
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spontaneous bacterial peritonitis: cirrhotic patients diagnosed with SBP
  Interventions: Diagnostic Test: ASCITIC FLUID CULTURE
- spontaneous fungal peritonitis: irrhotic patients diagnosed with SFP
  Interventions: Diagnostic Test: ASCITIC FLUID CULTURE

INTERVENTIONS:
Diagnostic Test: ASCITIC FLUID CULTURE — Ten milliliters of ascitic fluid will be collected at the bedside and inoculated into aerobic and anaerobic blood culture bottles. Bacterial culture will be performed manually using MacConkey and blood agar plate

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is an infection of the peritoneal cavity with no surgically treatable intra-abdominal source of infection. Spontaneous peritonitis is a potentially fatal complication in patients with advanced liver cirrhosis. It is estimated that 10-20 % of patients with cirrhotic ascites may develop spontaneous peritonitis, which is usually caused by a bacterial infection.

In contrast, spontaneous fungal peritonitis (SFP) is less well-recognized. SFP may be associated with higher mortality rates than SBP but therapeutic approaches are largely undefined. To this end, the epidemiology and outcomes of patients with SFP have only been documented sporadically aimed to evaluate the risk factors for the development of spontaneous fungal peritonitis (SFP), and the prognosis of SFP compared with SBP

DETAILED DESCRIPTION:
Cross-sectional study

Studied population & locality:

Patients with signs and symptoms suggestive of spontaneous peritonitis who will be admitted to Tropical medicine and Gastroenterology or Internal medicine departments in Sohag university hospitals during the period from september 2021 to december 2022 will be included in the study.

According to the results of ascitic fluid analysis, we will divide the patients into 2 groups:

Group (1): patients with spontaneous bacterial peritonitis (SBP). Group (2): patients with spontaneous fungal peritonitis (SFP).

Exclusion criteria:

Patients seropositive for human immunodeficiency virus (HIV) and patients undergoing continuous ambulatory peritoneal dialysis were excluded from this study.

Methods:

All included patients will be subjected to:

1. Detailed history, complete general and systemic examination.
2. Ascitic fluid analysis
3. Bacterial and fungal culture from ascitic fluid:
4. Laboratory investigations:

Fasting blood sugar Liver function tests. CBC.

Ethical considerations:

ELIGIBILITY:
Inclusion Criteria:

Patients with signs and symptoms suggestive of spontaneous peritonitis who will be admitted to Tropical medicine and Gastroenterology or Internal medicine departments in Sohag university hospitals during the period from September 2021 to december 2022

Exclusion Criteria:

Patients seropositive for human immunodeficiency virus (HIV) and patients undergoing continuous ambulatory peritoneal dialysis were excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with signs and symptoms suggestive of spontaneous peritonitis who will be admitted to Tropical medicine and Gastroenterology or Internal medicine departments in Sohag university hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
he risk factors for the development of spontaneous fungal peritonitis | September 2021 to December 2022 will be included in the study.
  number/percentage

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Farag, MD, Study Chair — Sohag University; osamaa orabi, MD, Study Chair — Sohag University
Locations (1):
- Mona Mohammed Abdelrahman, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang SY, Yu SJ, Lee JH, Kim JS, Yoon JW, Kim YJ, Yoon JH, Kim EC, Lee HS. Spontaneous fungal peritonitis: a severe complication in patients with advanced liver cirrhosis. Eur J Clin Microbiol Infect Dis. 2014 Feb;33(2):259-64. doi: 10.1007/s10096-013-1953-2. Epub 2013 Sep 2. PMID 23996048
- [Background] Bremmer DN, Garavaglia JM, Shields RK. Spontaneous fungal peritonitis: a devastating complication of cirrhosis. Mycoses. 2015 Jul;58(7):387-93. doi: 10.1111/myc.12321. Epub 2015 Apr 7. PMID 25851525
- [Background] Shizuma T. Spontaneous bacterial and fungal peritonitis in patients with liver cirrhosis: A literature review. World J Hepatol. 2018 Feb 27;10(2):254-266. doi: 10.4254/wjh.v10.i2.254. PMID 29527261